CLINICAL TRIAL: NCT01492153
Title: A Post Marketing Surveillance on the Use of NovoLet® Human Insulin System in Indonesia
Brief Title: NovoLet® Surveillance Study on Using Human Insulin System in Indonesia
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NOPEN3-1886
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — biphasic human insulin 30; Insulin, Isophane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NovoLet® device
  Interventions: Drug: biphasic human insulin; Drug: isophane human insulin; Drug: human soluble insulin

INTERVENTIONS:
Drug: biphasic human insulin — NovoLet® device delivering human insulin. Selection of drug and timing of dose for each patient was at the discretion of the investigator
Drug: isophane human insulin — NovoLet® device delivering human insulin. Selection of drug and timing of dose for each patient was at the discretion of the investigator
Drug: human soluble insulin — NovoLet® device delivering human insulin. Selection of drug and timing of dose for each patient was at the discretion of the investigator

SUMMARY:
This study is conducted in Asia. The aim of this study is to investigate the safety and efficacy of NovoLet® human insulin delivery system in an outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus
* Type 2 diabetes mellitus
* Other types of diabetes mellitus (gestational, drug induced [thiazide] or metabolic syndrome-related)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 1 or type 2 diabetes mellitus or other types of diabetes mellitus (gestational, drug induced or metabolic syndrome-related) who are prescribed NovoLet® human insulin in the course of their diabetes mellitus management can be enrolled in the study
Sampling Method: Probability Sample
Enrollment: 1981 (Actual)
Dates: Start 2003-02-11 (Actual); Primary Completion 2006-09-05 (Actual); Study Completion 2006-09-05 (Actual)

PRIMARY OUTCOMES:
Change in body weight

SECONDARY OUTCOMES:
Fasting blood glucose (FBG)
2 hours postprandial blood glucose (2-hr PPBG)
HbA1c (glycosylated haemoglobin)
Adverse events (AEs) including hypoglycaemic episodes

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1457), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Jakarta, Indonesia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com